CLINICAL TRIAL: NCT06632119
Title: Immediate Effects of High-intensity Laser Therapy on Knee Joint Position Sense and Knee Muscle Strength in Patients with Knee Osteoarthritis
Acronym: HILT on KOA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Prasert Sakulsriprasert, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU_CIRB 2024/003.0401
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: HILT; Laser therapy; joint sense; muscle strength; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HILT (Active Comparator): high-intensity laser therapy (HILT)
  Interventions: Device: high-intensity laser therapy
- Sham_HILT (Placebo Comparator): Sham-HILT, the HILT without laser release
  Interventions: Device: Sham-HILT

INTERVENTIONS:
Device: high-intensity laser therapy — high-intensity laser therapy (HILT) machine, ASA laser
  Arms: HILT
Device: Sham-HILT — Sham-HILT, HILT machine without laser release
  Arms: Sham_HILT

SUMMARY:
The goal of this clinical trial is to compare whether HILT versus Sham-HILT is effective to reduce pain, improve knee joint position sense, and knee muscle strength.

Participants will undergo a single-session of HILT or Sham-HILT, the measurements of pain, knee joint position sense error, and knee muscle strength will be done at before, immediately after, and 24-hour after the single-session intervention.

DETAILED DESCRIPTION:
The investigators would like to investigate whether single session of high-intensity laser therapy (HILT) is promising to see the changes in individuals with knee osteoarthritis (KOA)-related knee pain regarding pain intensity, knee joint position sense, and knee muscle strength.

The objectives of this study is to compare pre and post, and between the two groups (HILT versus Sham-HILT) at after interventions regarding pain, knee joint position sense, and knee muscle strength.

Participants will undergo a single-session of HILT or Sham-HILT by an experienced musculoskeletal physical therapist, the measurements of pain, knee joint position sense error, and knee muscle strength will be done at before, immediately after, and 24-hour after the single-session intervention.

ELIGIBILITY:
Inclusion Criteria:

* knee pain greater than 3 on the Visual Analog Scale (VAS) for more than 3 months
* diagnosed with unilateral knee osteoarthritis by a physician or meeting the American College of Rheumatology Classification Criteria for clinical knee osteoarthritis
* the severity of knee osteoarthritis is classified as grades 0-3 according to the Kellgren-Lawrence (KL) classification
* should not have undergone any specific treatments in the 3 months preceding the recruitment for the study, such as steroid injections.

Exclusion Criteria:

* any other musculoskeletal problems associated with knee pain
* musculoskeletal problems associated with the hip and ankle joints
* a history of lower limb fracture
* neurological conditions
* contraindications for laser therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Knee joint position sense | Baseline, immediately after, 24-hour after intervention
  Knee joint position sense, the investigators used the joint position repositioning technique. The participants were measured for joint position reposition technique with a smartphone application "Measure App" (iPhone 12 Pro Max, Apple Inc., USA). The smartphone attached at shank of tibia bone at the malleolar level. The participants sat in the starting position knee flexion 90°. Then the participants with eyes closed were actively guided to the knee flexion 45 degrees and hold for 3 seconds. The data was recorded the difference between performed position and targeted position.

SECONDARY OUTCOMES:
Knee muscle strength | Baseline, immediately after, 24-hour after intervention
  The muscle strength measured both quadriceps and hamstring muscles by the handheld dynamometer at 90°.
Pain | Baseline, immediately after, 24-hour after intervention
  The participants rated the pain scores using a 10-cm visual analog scale (VAS) ranged from 0 "no pain at all" on the left end to 10 "worst pain imaginable" on the right end.

CONTACTS AND LOCATIONS:
Overall Officials: Prasert Sakulsriprasert, Ph.D., Principal Investigator — Mahidol University
Locations (1):
- Physical Therapy, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No
This is a pilot study